CLINICAL TRIAL: NCT00935142
Title: Non Invasive Imaging of [18F]VM4-037 With Positron-Emission-Tomography (PET): A Phase I Trial
Brief Title: Non-invasive Imaging With [18F]VM4-037
Acronym: [18F]VM4-037
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: [18F]VM4-037; CaIX
Record Dates: First submitted 2009-06-30; First posted 2009-07-08 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Stage 4 Cancer
Keywords: stage IV cancer with no treatment options; non-curative
MeSH Terms: conditions — Neoplasms | interventions — 3-(4-(2-fluoroethoxy)phenyl)-2-(3-methyl-2-(4-((2-sulfamoylbenzo(d)thiazol-6-yloxy)methyl)-1H-1,2,3-triazol-1-yl)butanamido)propanoic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: [18F]VM4-037 — Bolus IV injection of [18F]VM4-037

SUMMARY:
The purpose of this study is to determine the toxicity of the hypoxia PET-tracer [18F]-VM4-037 in cancer patients in two dose-steps:

* Step 1 (3-6 patients): a single dose of maximum 8 mCi (296 MBq) dose of [18F]VM4-037 via a bolus IV injection.
* Step 2 (3-6 patients): a single dose of maximum 12 mCi (444 MBq) dose of [18F]VM4-037 via a bolus IV injection

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmed solid tumour, primary or secondary stage IV and/ or tumours with no curative treatment options
* WHO performance status 0 to 1
* Normal white blood cell count and formula
* Normal platelet count
* No anaemia requiring blood transfusion or erythropoietin
* Adequate hepatic function: Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for the institution; ALT, AST, and alkaline phosphatase ≤ 2.5 x ULN for the institution)
* Calculated Creatinin clearance at least 60 ml/min
* No administration of Fluor-18 in the previous 24 hours
* The patient is capable of complying with study procedures
* 18 years or older

Exclusion Criteria:

* Only visible tumor sites in the upper abdomen (because the uptake of VM4-037 in the liver, stomach and the kidneys would interfere with image quality of the tumor)
* Known hypersensitivity for sulfonamides
* Recent (< 3 months) myocardial infarction
* Uncontrolled infectious disease
* Less than 18 years old
* Pregnancy
* No concurrent anti-cancer agents or radiotherapy allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Toxicity (CTCAE 3.0) | 1 week

SECONDARY OUTCOMES:
Image Quality | 1 week
Correlation with circulating biomarkers of hypoxia | 1 week
Correlation with [18F]-FDG on PET scans | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, MD. PhD., Principal Investigator — Maastro Clinic, The Netherlands